CLINICAL TRIAL: NCT06645652
Title: Feasibility and Preliminary Effects of a Drawing-based Intervention on Cognition and Wellbeing of Community-Dwelling Adults at Risk for ADRD
Brief Title: Visual Arts Interventions With Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NU-DS-20241011
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Feasibility Study
Keywords: Cognition; Perception; Aged; Healthy Volunteers; Learning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participatory Arts (Experimental): Participants will develop drawing skills through learning specific techniques and deliberately engaging cognitive domains such as perception, visuospatial reasoning, attention, and processing speed. The intervention is completed in a hybrid format where lessons are completed online and practice is completed in a sketchbook and drawing things from life. Prompts are provided to guide daily practice sessions. Techniques learned include contour drawing, gesture drawing, negative space drawing.
  Interventions: Behavioral: Training in observational drawing
- Receptive Arts (Active Comparator): Participants will learn about different art periods and browse online galleries. The materials will be available online through a website through which participants will access and browse online galleries. Weekly topics include genres, subjects, or specific mediums. Prompts and vocabulary will accompany the galleries to guide their learning.
  Interventions: Behavioral: Arts engagement through digital galleries

INTERVENTIONS:
Behavioral: Training in observational drawing — * 6 weeks of online gallery browsing based on different topics
  * Daily practice drawing from observation with training adding up to 1 hour a week
  * Documenting progress and reflection writing
  Arms: Participatory Arts
Behavioral: Arts engagement through digital galleries — * 6 weeks of online gallery browsing based on different topics
  * 2 hours of weekly activities consist of reading and navigating technology
  * Reflection writing
  Arms: Receptive Arts

SUMMARY:
The present study investigates the feasibility, acceptability, and preliminary effects of a novel visual arts-based intervention in an older adult population. In a randomized controlled design, two arts-based interventions will be evaluated with a group of 50 participants.

DETAILED DESCRIPTION:
A two-arm randomized controlled study will be conducted to obtain within-group ratings of feasibility and acceptability, as well as between-group differences in drawing skills after training. In the drawing intervention, participants will learn and train drawing skills through exercises that target attention, perception, and visuospatial reasoning. In the active control condition, participants will navigate virtual art galleries. Both interventions will be completed remotely and at home. Participants will complete in-lab assessment sessions before and after the training.

Each intervention consists of 6 weeks of training for up to 2 hours a week, including up to 1 hour of a self-guided lesson and prompted daily drawing practice adding up to 1 hour in the drawing intervention and 2 1-hour sessions of virtual gallery exploring per week in the arts appreciation intervention. The pre-test is administered within one week of the start of training and the post-test is administered within one week of training completion.

ELIGIBILITY:
Inclusion Criteria:

* 55-85 years of age
* Able to understand and speak English and follow study procedures
* Does not have a psychological or neurological condition that would prevent from being able to give consent to participate
* Less than 2 years of formal visual arts training

Exclusion Criteria:

* Formal diagnosis of dementia or other neurological disease, including Mild Cognitive Impairment
* A final score below 17 on the Montreal Cognitive Assessment - Blind (phone) version
* Abnormal visual acuity prohibitive of tablet-based training
* Physical handicap (motor or perceptual) that would impede training procedures
* Medical illness requiring treatment and/or significant absences during the study timeline

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability - clarity | Throughout training and post-test 6-8 weeks later
  Perceived clarity on the course content, likert scale 1-5
Acceptability - engagement | Throughout training and post-test 6-8 weeks later
  Level of engagement with the course materials, likert scale 1-5
Acceptability - value | Throughout training and post-test 6-8 weeks later
  Perceived value of the course content, likert scale 1-5
Feasibility - completion rate | Throughout training and post-test 6-8 weeks later
  % of participants who completed both testing sessions
Feasibility - adherence | Throughout training and post-test 6-8 weeks later
  % of lessons that participants completed, from 0-6
Feasibility - frequency | Throughout training and post-test 6-8 weeks later
  Frequency: times a week that participants completed training, 0-7 for days practiced each week
Feasibility - attrition | Throughout training and post-test 6-8 weeks later
  Attrition reason: participants withdrawing will select from one of 5 options or 'other' to record the reason for withdrawing
Change in Drawing skills | Pre-test (baseline) and post-test 6-8 weeks later
  Participants will have 5 minutes to draw a photograph. Accuracy is scored using two methods: angle error at defined points of intersection and a rubric assessing accuracy on global and local features. Both ratings are averaged into a composite z-score, as well as looked at separately.

SECONDARY OUTCOMES:
Change in Perception - contour integration | Pre-test (baseline) and post-test 6-8 weeks later
  Participants tap on circles of aligned Gabors embedded in a scene of randomly oriented Gabors. A circle will be present for 3 seconds and switch to the next trial if it is not seen. Number of circles spotted, reaction times on spotted circle, and lowest level of alignment will be recorded. Z-scores will be calculated.
Change in Perception - visual disembedding | Pre-test (baseline) and post-test 6-8 weeks later
  Participants search for a target shape in 3 complex gestalts of overlapping shapes. Participants select the complex shape containing the target. Response times and accuracy are measured. Z-scores will be calculated.
Change in Visuospatial Reasoning - construction and memory | Pre-test (baseline) and post-test 6-8 weeks later
  Complex Figures Copy and Recall will assess visuospatial construction and memory (10 min). Participants will complete three sets of drawing complex shapes from observation and memory after a block of word learning. Accuracy will be scored using a validated rubric.
Change in Visuospatial Reasoning - mental transformation | Pre-test (baseline) and post-test 6-8 weeks later
  3D Mental Rotation (3 min) will test mental transformation. Participants will be briefly shown two figures and asked to determine whether the figures are the same or mirror reversed. Mean and SD reaction time per angular disparity and errors per angular disparity will be extracted.
Change in Attention | Pre-test (baseline) and post-test 6-8 weeks later
  A Rule switch task will measure set shifting. Participants will sort shapes by color or shape. Performance will be calculated as the response times on accurate switch trials.
Change in Mindfulness | Pre-test (baseline) and post-test 6-8 weeks later
  Participants complete a version Solloway Mindfulness Survey adapted to drawing. The questionnaire includes 30 questions on a 7-point scale on the degree to which engaging in drawing is related to different aspects of mindful attention.
Change in Mental Wellbeing | Pre-test (baseline) and post-test 6-8 weeks later
  Mental Wellbeing is assessed by the WEMWBS, which includes 14 questions on a 5 point scale about positive mental wellbeing.

OTHER OUTCOMES:
Daily progress log | After every training session (weeks 1-6 of training, up to 7 times a week)
  Participants will record the time spent and the content practiced during their sessions. The survey includes selecting all the choices that apply, questions on a likert scale, and short response questions.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Jaeggi, PhD, Principal Investigator — Northeastern University; Aaron Seitz, PhD, Principal Investigator — Northeastern University

IPD SHARING:
Plan to Share IPD: Yes
Intervention materials and individual participant data (anonymized)
Supporting Information: Study Protocol
Time Frame: Data will be available persistently at the conclusion of the study.
Access Criteria: There are no access criteria.